CLINICAL TRIAL: NCT06821100
Title: Thymalfasin (Thymosin Alpha 1; Ta1) as an Enhancer of Vaccine Response Among Older Adults Receiving Booster Doses of COVID-19 Vaccine
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00037612
Record Dates: First submitted 2025-01-15; First posted 2025-02-11 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Vaccine Response; COVID-19 Vaccine; Immune Response to Covid 19 Vaccination
MeSH Terms: interventions — Thymalfasin; Trace amine-associated receptor 1

STUDY DESIGN:
Intervention Model Description: A randomized open label Phase 1 study to evaluate the safety and tolerability of different treatment regimens of Ta1 before vaccination with a SARS-CoV-2 mRNA vaccine. Study participants will be randomized in a 1:1:1 ratio to one of the following treatment groups:
  * No Ta1 prior to vaccination (Control)
  * A 4.8 mg dose of Ta1 (dose of 1.6 mg in 1 mL of diluent X3) on Day 0, followed by vaccination (Treatment arm A)
  * A 4.8 mg dose of Ta1 (dose of 1.6 mg in 1 mL of diluent X3) on Day 0 and Day 3, followed by vaccination (Treatment arm B)
  * All participants will receive the same mRNA SARS-CoV-2 mRNA vaccine (Moderna or Pfizer) for consistency.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): No Ta1 prior to vaccination
- Treatment arm A (Experimental): A 4.8 mg dose of Ta1 (dose of 1.6 mg in 1 mL of diluent X3) on Day 0, followed by vaccination
  Interventions: Drug: Thymalfasin (Thymosin alpha 1, Ta1)
- Treatment arm B (Experimental): A 4.8 mg dose of Ta1 (dose of 1.6 mg in 1 mL of diluent X3) on Day 0 and Day 3, followed by vaccination
  Interventions: Drug: Thymalfasin (Thymosin alpha 1, Ta1)

INTERVENTIONS:
Drug: Thymalfasin (Thymosin alpha 1, Ta1) — Ta1 is a naturally occurring peptide that has been evaluated for its immunomodulatory activities and related therapeutic potential in several conditions and diseases. Ta1 has been shown to provide increased response to vaccines.
  Arms: Treatment arm A; Treatment arm B

SUMMARY:
The goal of this research is to learn more about ZADAXIN® (trade name; thymalfasin generic; Ta1 for short) and determine if Ta1 has any benefit in increasing the immune response to the COVID-19 vaccine. Ta1 has been shown to stimulate the immune system to fight infections.

This research study will test the safety and possible harms of Ta1 when it is given to people at different dose levels before COVID-19 vaccination.

ELIGIBILITY:
Inclusion Criteria

Subjects who meet all of the following criteria will be eligible to participate in the study:

1. Age 65 or greater.
2. Able and willing to provide informed consent or have consent provided by a legally authorized representative (LAR).
3. Scheduled for SARS-CoV-2 mRNA vaccination booster dose.
4. If a male subject, the subject must agree to use barrier contraception (ie, condoms) from Day 1 through 30 days following the last dose of study drug.

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from participation in the study.

Laboratory related exclusion criteria should be assessed using historical records and lab results available in the subjects' electronic medical records.

1. Hypoxemia for any reason, defined as either oxygen saturation (SpO2) ≤ 93% on room air or a requirement for supplemental oxygen support.
2. Participants with one of the following:

   * Acute liver failure defined as INR ≥ 1.5 and altered mental status in a patient without cirrhosis or pre-existing liver disease.
   * Acute kidney failure defined as an increase in serum creatinine of ≥0.3 mg/dL within 48 hours or ≥50% within 7 days OR urine output of <0.5 mL/kg/hour for >6 hours
   * Heart failure with NYHA functional classification III or IV.
3. Advanced cancer being treated with cytotoxic chemotherapy.
4. Participants have end stage renal disease requiring hemodialysis or peritoneal dialysis, or chronic kidney disease with GFR < 30 mL/min/1.73m2
5. Participants with a known history of cirrhosis and Child-Pugh score B or C.
6. Participants who are moderately or severely immunocompromised defined as:

   * Are receiving active treatment for solid tumor and hematologic malignancies.
   * Have hematologic malignancies (e.g., chronic lymphocytic lymphoma, non-Hodgkin lymphoma, multiple myeloma, acute leukemia) and are known to have poor responses to COVID-19 vaccines, regardless of the treatment status for the hematologic malignancy.

   Received a solid-organ or islet transplant and are receiving immunosuppressive therapy.
   * Received chimeric antigen receptor T cell (CAR T-cell) therapy or a hematopoietic cell transplant (HCT) and are within 2 years of transplantation or are receiving immunosuppressive therapy.
   * Have a moderate or severe primary immunodeficiency (e.g., severe combined immunodeficiency, DiGeorge syndrome, Wiskott-Aldrich syndrome, common variable immunodeficiency disease).
   * Have advanced or untreated HIV infection (defined as people with HIV and CD4 T lymphocyte cell counts <200 cells/mm3, a history of an AIDS-defining illness without immune reconstitution, or clinical manifestations of symptomatic HIV).
   * Are receiving active treatment with high-dose corticosteroids (i.e., ≥20 mg prednisone or equivalent per day for ≥2 weeks), alkylating agents, antimetabolites, transplant-related immunosuppressive drugs, cancer chemotherapeutic agents classified as severely immunosuppressive, or immunosuppressive or immunomodulatory biologic agents (e.g., B cell-depleting agents).
7. Participants with uncontrolled autoimmune or rheumatologic disease.
8. Participants have received 6 doses or more of the COVID-19 vaccine. (Removed in Amendment 3)
9. Participants with a history of myocarditis, pericarditis, or myopericarditis.
10. Participants with a history of anemia or bleeding disorders. For anemia, the exclusion criterion will be met if any of the following are true:

    i. Active anemia, defined as Hb<9 g/dL within 30 days prior to screening,

    ii. Unresolved anemia: Hb<11 g/dL (females) or <12 g/dL (males) during any window of >=3 months in the past year AND no evidence of measures of correction (e.g. iron supplementation, transfusion) in the same time window,

    iii. High risk etiologies of anemia: myelodysplastic syndromes, aplastic anemia, hemoglobinopathies (e.g., sickle cell trait, sickle cell anemia), anemia due to malignancy, anemia due to chronic kidney disease, anemia due to untreated nutritional deficiencies, anemia due to toxic exposures (e.g., chronic lead poisoning), or any other high-risk etiology as determined by the study investigator,

    iv. Anemia with intensive recent (within 6 months) interventions, including red blood cell transfusion or IV iron infusion,

    v. Symptomatic anemia in the year prior to screening, including shortness of breath, exercise intolerance, type 3 myocardial infarction, if clearly attributed to the anemia.
11. Participants who have precautions or contraindications to COVID-19 vaccine per the CDC interim clinical considerations for use of COVID-19 vaccines, including the following:

    * History of a severe allergic reaction (e.g., anaphylaxis) after a previous dose or to a component of the COVID-19 vaccine
    * History of a diagnosed non-severe allergy to a component of the COVID-19 vaccine
    * History of a non-severe, immediate (onset less than 4 hours) allergic reaction after administration of a previous dose of one COVID-19 vaccine type
    * Moderate or severe acute illness, with or without fever
    * History of multisystem inflammatory syndrome in adults
    * History of myocarditis or pericarditis within 3 weeks after a dose of any COVID-19 vaccine
12. History of allergy or intolerance to Ta1.
13. SARS-CoV-2 or other infection, during screening.
14. SARS-CoV-2 mRNA or other SARS-CoV-2 vaccination during the previous 6 months.
15. Participants who have dermatologic conditions that could affect local solicited adverse event (AE) assessment (e.g., psoriasis patches affecting skin over the sites of injection).
16. Any medical condition that, in the judgement of the Investigator, could interfere with treatment or compliance with the protocol.
17. Has received an investigational drug within the previous 30 days.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 52 weeks
  The primary objective is to evaluate the safety and tolerability of different treatment regimens of Ta1 before vaccination with a SARS-CoV-2 mRNA vaccine. This will be measured by:
  - The incidence and severity of adverse events (AEs) following treatment

SECONDARY OUTCOMES:
Levels of neutralizing and non-neutralizing antibodies | 24 weeks
  Levels of neutralizing and non-neutralizing antibodies. Data will be summarized descriptively for each treatment arm and no formal hypothesis testing is planned
Neutralizing activity to SARS-CoV-2 | 24 weeks
  Neutralizing activity to SARS-CoV-2, measured using a using a pseudovirus neutralization assay. Data will be summarized descriptively for each treatment arm and no formal hypothesis testing is planned
T cell response | 24 weeks
  T cell response. Data will be summarized descriptively for each treatment arm and no formal hypothesis testing is planne

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No